CLINICAL TRIAL: NCT00925938
Title: A Phase II, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging Study to Assess the Efficacy and Safety of the Misoprostol Vaginal Priming Insert for Women Requiring Cervical Priming Prior to a Hysteroscopy
Brief Title: Efficacy and Safety Study of the Misoprostol Vaginal Priming Insert (MVPI) Prior to Hysteroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Miso-Gyn-201
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Cervical Priming
Keywords: Hysteroscopy; Cervical priming; Cervical dilatation; Misoprostol; Endoscopy, uterine
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol vaginal priming insert (MVPI) (Experimental): One vaginal insert administered 18 - 24 hours prior to the scheduled hysteroscopy clinic visit. The initial dose is 400 mcg and dose will be adjusted between 100 - 1600 mcg after each study cohort based on safety and efficacy criteria as assessed by the Data and Safety Monitoring Board (DSMB).
  Interventions: Drug: misoprostol
- MVPI Placebo (Placebo Comparator): One vaginal insert of placebo administered 18 - 24 hours prior to the scheduled hysteroscopy clinic visit.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: misoprostol — One vaginal insert containing 100, 200, 400, 800, 1200, 1600 mcg misoprostol administered intravaginally one time and remain in place for 18 - 24 hours prior to the hysteroscopy procedure. An adaptive design will be used to determine whether to escalate or reduce the dose, starting with MVPI 400 mcg.
  Arms: Misoprostol vaginal priming insert (MVPI)
Drug: placebo — placebo
  Arms: MVPI Placebo

SUMMARY:
A Phase II, multicenter, double-blind, randomized, placebo-controlled, dose-ranging, study to assess the efficacy and safety of the 100, 200, 400, 800, 1200 and 1600 mcg Misoprostol Vaginal Priming Insert (MVPI) for Women Requiring Cervical Priming prior to an in-office hysteroscopy procedure. Each subject will be randomized to receive one vaginal insert. The study drug will be administered vaginally by a member of the clinical research team (Part I) or insert herself (Part II) 18 - 24 hours prior to the scheduled hysteroscopy clinic visit. The internal os of the cervix will be measured at baseline, just prior to the hysteroscopy and at the follow up visit. The primary outcome measure is change in diameter of the internal cervical os from baseline (pre-treatment) to just prior to the hysteroscopy procedure (post-treatment). The hypothesis is that treatment with the MVPI will soften and dilate the cervix better than placebo.

DETAILED DESCRIPTION:
Prior to the hysteroscopy procedure, study staff will record the type of procedure that will be conducted and the desired cervical dilatation. The study drug will be removed in the office and then a vaginal examination will be performed for signs of irritation or trauma. The diameter of the internal os will then be assessed using Hegar dilators. The diameter of the internal os will be assessed by the largest size of Hegar dilator that can be inserted into the internal os without resistance. If the subject requires further dilatation prior to the procedure, this will be noted; additional dilatation is per clinician preference. The use of a tenaculum to allow insertion of the dilator(s)/ hysteroscope should be recorded. The time of starting and ending the hysteroscopy procedure will be documented. The start time of the hysteroscopy procedure is taken from the time of insertion of the first Hegar dilator to completion of the hysteroscopy procedure. Cervical priming assessment and safety will be recorded.

The subject will attend the clinic for follow-up assessments 7 days after the procedure.

Adverse events and concomitant medications will be recorded throughout the study.

The study will use an adaptive design, beginning with the MVPI 400 mcg and escalating or reducing the dose depending on results seen with a particular dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, pre-menopausal women;
* Women aged 18 years and above;
* Women who are undergoing an in-office procedure requiring uterine access along with a cervical dilatation of at least 5.5 mm;
* Women participating in Part 1 of study: Women who have had at least one vaginal delivery of at least 24 weeks gestation;
* Women with Pap smear results that do not require further evaluation for at least one year as assessed by the investigator. Note: 1) results must be from a Pap smear obtained within one year of screening; 2) if results are unavailable or not current, a Pap smear must be obtained and results reviewed prior to study inclusion; 3) if a Pap smear is to be performed at screening, subject must have a negative pregnancy test confirmed prior to the Pap smear collection;
* Women of child bearing potential: 1) Must have a negative urine pregnancy test at screening and just prior to study drug insertion, if this takes place on a different day from the screening visit; 2) Agree to use a highly effective method of birth control (defined as a low failure rate of less than 1% per year) as follows: implants, injectables, combined oral contraceptives, sexual abstinence from the date of the subject's last menstruation until completion of the follow-up visit, vasectomised partner or barrier method (condom with spermicide). Women in a same sex relationship do not need to meet this criterion if they confirm that there is no possibility of pregnancy;
* Women who agree to refrain from vaginal intercourse while the study drug is in place;
* Women who agree to refrain from using any of the following from the day of study drug insertion until completion of the follow-up visit: feminine deodorant sprays/products, spermicides*, douches, condoms*, tampons, diaphragms or any other pharmaceutical or over the counter vaginal product. Barrier methods of contraception as indicated above (*) may be resumed following the dilatation procedure;
* Women who provide written informed consent.

Exclusion Criteria:

* Menopausal women;
* Women with menstrual periods lasting >10 days in duration;
* Baseline internal cervical os ≥ 3 mm;
* Women who have had prior endometrial ablation;
* Women who are breastfeeding;
* History or current diagnosis of glaucoma;
* Women with clinically significant vaginal or cervical abnormality (e.g. symptoms of an infection) that would interfere with conducting study procedures prior to study drug insertion;
* Women who are currently undergoing treatment for cancer (basal cell carcinoma is acceptable);
* Body Mass Index (BMI) ≥ 50;
* Women participating in Part 1 of study: Women with a history of loop electrosurgical excision procedure (LEEP) or cold knife conization without an intervening vaginal delivery;
* Women with an intra-uterine device (IUD) in place, had an IUD removed within 30 days of the screening visit or scheduled to have an IUD inserted during the hysteroscopy procedure;
* Women using NuvaRing® for contraception;
* Known or suspected allergy to misoprostol, other prostaglandins or any of the excipients;
* Unable to comply with the protocol.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (2):
- United States (2):
  - Precision Trials, Phoenix, Arizona
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Premenopausal women requiring cervical priming prior to an in-office hysterectomy procedure were recruited at 5 sites in the US
Pre-assignment Details: Part 1 of the study included only women who had at least one vaginal delivery. There was no restriction on vaginal delivery status in Part 2 of the study.
  Part 1 participants were included in the MVPI 400 mcg cohort, MVPI 800 mcg cohort and the Placebo cohort.
  Part 2 participants were included in the MVPI 800 mcg cohort and the Placebo cohort.
Groups:
- MVPI 400 Mcg: One vaginal insert administered 18 - 24 hours prior to the scheduled hysteroscopy clinic visit.
  Part 1 participants were included in this arm of the study.
  misoprostol : One vaginal insert containing 400 mcg misoprostol administered intravaginally one time and remain in place for 18 - 24 hours prior to the hysteroscopy procedure.
- MVPI 800 Mcg: One vaginal insert administered 18 - 24 hours prior to the scheduled hysteroscopy clinic visit.
  Part 1 and Part 2 participants were included in this arm of the study.
  Following the initial dose, 400 mcg, the dose was increased to 800 mcg after the 400 mcg group cohort based on safety and efficacy criteria as assessed by the Data and Safety Monitoring Board (DSMB).
- MVPI Placebo: One vaginal insert of placebo administered 18 - 24 hours prior to the scheduled hysteroscopy clinic visit.
  Part 1 and Part 2 participants were included in this arm of the study.
  placebo : placebo
Period: Overall Study
Arm/Group | MVPI 400 Mcg | MVPI 800 Mcg | MVPI Placebo
Started | 9 | 25 | 17
Completed | 9 | 25 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MVPI 800 Mcg: One vaginal insert administered 18 - 24 hours prior to the scheduled hysteroscopy clinic visit. Following the initial dose, 400 mcg, the dose was increased to 800 mcg after the 400 mcg group cohort based on safety and efficacy criteria as assessed by the Data and Safety Monitoring Board (DSMB). Part 1 and Part 2 participants were included in this arm of the study.
- Total: Total of all reporting groups
Arm/Group | MVPI 400 Mcg | MVPI 800 Mcg | MVPI Placebo | Total
Number analyzed (Participants) | 9 | 25 | 17 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 25 | 17 | 51
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (6.57) | 41.5 (6.21) | 42.0 (5.86) | 41.5 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 25 | 17 | 51
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 25 | 17 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change in Diameter of the Internal Cervical os From Baseline (Pre-treatment) to Just Prior to the Hysteroscopy Procedure (Post-treatment).
Time Frame: Baseline to 18-24 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MVPI 400 Mcg | MVPI 800 Mcg | MVPI Placebo
Number analyzed (Participants) | 9 | 25 | 17
mm | 2.2 (1.86) | 2.3 (2.21) | 1.5 (1.84)

2. Secondary Outcome: Percent of Women Requiring Further Dilatation in Order to Allow Uterine Access
Time Frame: 18 - 24 hours
Population: A total of 46 subjects (90.2%) did not achieve their target dilatation after study drug removal (MVPI 400: 8 subjects; MVPI 800: 21 subjects; Placebo: 17 subjects). Forty-five subjects had additional dilatation attempted; additional dilatation was not attempted on one subject (MVPI 800) due to a protocol deviation (MVPI 800: 20 subjects).
Measure: Number; unit: percentage of participants
Arm/Group | MVPI 400 Mcg | MVPI 800 Mcg | MVPI Placebo
Number analyzed (Participants) | 9 | 25 | 17
percentage of participants
  Subjects requring additional dilatation | 88.9 | 84.0 | 100
  Target Dilation Achieved following 2ndry dilation | 100 | 85.0 | 100

3. Secondary Outcome: Total Procedure Time From Insertion of the First Hegar Dilator to Completion of the Hysteroscopy Procedure;
Time Frame: 18 - 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | MVPI 400 Mcg | MVPI 800 Mcg | MVPI Placebo
Number analyzed (Participants) | 9 | 25 | 17
minutes | 3.26 (3.931) | 3.75 (5.888) | 2.32 (1.573)

4. Secondary Outcome: Physician Assessment of Ease of Cervical Dilation;
Time Frame: 18 - 24 hours
Measure: Number; unit: percentage of participants
Arm/Group | MVPI 400 Mcg | MVPI 800 Mcg | MVPI Placebo
Number analyzed (Participants) | 9 | 25 | 17
percentage of participants
  Inadequate | 22.2 | 36.0 | 47.1
  Adequate/ Correct Softness | 66.7 | 48.0 | 52.9
  Over Primed/ Too soft | 11.1 | 16.0 | 0

5. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: 9 days
Measure: Number; unit: Percentage of participants
Arm/Group | MVPI 400 Mcg | MVPI 800 Mcg | MVPI Placebo
Number analyzed (Participants) | 9 | 25 | 17
Percentage of participants | 100 | 92.0 | 82.4

ADVERSE EVENTS:
Time Frame: All AEs were followed until resolution,the condition stabilized or for at least 30 days after d/c of the study drug, whichever came first. All AEs that were reported spontaneously up to 2 weeks after the subject completed the study were recorded.
Arm/Group | MVPI 400 Mcg | MVPI 800 Mcg | MVPI Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/25 | 0/17
Other Adverse Events (participants affected / at risk) | 9/9 | 23/25 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVPI 400 Mcg (N=9) | MVPI 800 Mcg (N=25) | MVPI Placebo (N=17)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVPI 400 Mcg (N=9) | MVPI 800 Mcg (N=25) | MVPI Placebo (N=17)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 8 (9) | 19 (25) | 10 (10)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 4 (4) | 6 (6) | 3 (3)
Uterine spasm (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications resulting from the clinical trial must be in a form that does not reveal technical information that the Sponsor considers confidential or proprietary. A copy of any abstract, presentation or manuscript proposed for publication must be submitted to the Sponsor for review at least 30 days before its submission. If deemed necessary for protection of proprietary information prior to patent filing, a further delay of 60 days is required before any publication is submitted.